CLINICAL TRIAL: NCT03131544
Title: MRI Guided Transrectal Prostate Laser Ablation for Benign Prostatic Hypertrophy (BPH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prostate Laser Center, PLLC (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Prostate Laser Center BPH 01
Record Dates: First submitted 2017-04-16; First posted 2017-04-27 (Actual); Results first posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: BPH; Prostate Hyperplasia; Urinary Frequency/Urgency
Keywords: BPH; Benign Prostatic Hypertrophy; MRI; Prostate; Lower Urinary Tract Symptoms; Nocturia; Incomplete bladder emptying
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms; Nocturia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- FLA for BPH Active Treatment (Experimental)
  Interventions: Device: MRI Guided Transrectal Periuretheral Transitional Zone Ablation

INTERVENTIONS:
Device: MRI Guided Transrectal Periuretheral Transitional Zone Ablation — Patients will undergo an MRI guided transrectal ablation of tissue within the periuretheral transitional zone.
  Other Names: Visualase

SUMMARY:
Over 100,000 BPH procedures are performed annually in the US. The purpose of this study is to evaluate the effectiveness of performing MRI guided transrectal laser ablation using a 980 nm laser (VisualaseTM by Medtronic, Inc., a Minnesota, U.S.A. company) to treat benign prostatic hypertrophy (BPH). The laser system will be used to necrotize urological soft tissue within the prostate under MRI guidance. This will be a single center, single arm prospective trial with an anticipated enrollment of 10 men. Patients who elect this treatment option and choose to be part of the study will be enrolled consecutively.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of lower urinary track symptoms (LUTS).
2. Prostate volume of 40 - 200 cc.
3. Men ≥ 45 years old.
4. IPSS ≥ 15.
5. BPH Impact Index ≥ 5.

Exclusion Criteria:

1. History of prostate or bladder cancer, pelvic radiation, untreated bladder stones, or findings suggestive of likely underlying prostate cancer.
2. Need to catheterize to relieve obstruction.
3. Daily use of incontinence materials/padding.
4. Neurogenic or hypotonic bladder, Parkinson's Disease, or a history of uncontrolled diabetes.
5. Prior interventional or surgical treatment of BPH.
6. Penile prosthesis.
7. Artificial urinary sphincter or collagen bladder injection.
8. Urethral stricture.
9. Bleeding disorder/coagulopathy.
10. Inability to refrain from blood thinners in the peri-procedural period.
11. Inability or chooses not to provide informed consent.
12. Any serious medical condition which would make proceeding to treatment unsafe.
13. Significant contraindication to MRI or gadolinium contrast.
14. Hip replacement.
15. Lack of a rectum.
16. Life expectancy of less than two years.
17. Unable or unwilling to complete all required questionnaires and follow-up assessments.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2020-05-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Prostate Laser Center, PLLC, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Harman AL, Toth R, Karamanian A. Magnetic Resonance Imaging-Guided Transrectal Prostate Laser Ablation for Benign Prostatic Hyperplasia. J Vasc Interv Radiol. 2023 Nov;34(11):2024-2028. doi: 10.1016/j.jvir.2023.07.015. Epub 2023 Jul 21. No abstract available. PMID 37481065
- See also: Related Info — https://www.ProstateLaserCenter.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All the procedures were performed between May 2017 and May 2018. All procedures were performed at a free-standing magnetic resonance imaging (MRI) center, and pre-procedure and post-procedure visits were completed in an outpatient office.
Groups:
- Focal Laser Ablation (FLA) for BPH Active Treatment: MRI Guided Transrectal Periuretheral Transitional Zone Ablation: Patients will undergo an MRI guided transrectal ablation of tissue within the periuretheral transitional zone.
Period: Overall Study
Arm/Group | Focal Laser Ablation (FLA) for BPH Active Treatment
Started | 10
Completed | 9
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | FLA for BPH Active Treatment
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10
Prostate volume [Mean (Standard Deviation); unit: cubic centimeters (cc)] — Prostate volume was calculated by measuring the length, width, and height of the prostate on MRI and using an ellipsoid volume calculation (Ellipsoid volume = L x W x H x π/6).
  cubic centimeters (cc) | 69.3 (31.0)
International Prostate Symptom Score (IPSS) [Mean (Standard Deviation); unit: points] | 26.3 (4.96)
International Prostate Symptom Score (IPSS) Quality of Life (QoL) [Mean (Standard Deviation); unit: points] | 5.1 (0.83)
Benign Prostatic Hyperplasia (BPH) Impact Index [Mean (Standard Deviation); unit: points] | 9.7 (1.9)
Sexual Health Inventory For Men (SHIM) [Mean (Standard Deviation); unit: points] | 20 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: International Prostate Symptom Score (IPSS) Change
Description: The IPSS survey rates lower urinary tract symptom severity from 0 (none) to 35 (severe).
Time Frame: From baseline to 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Focal Laser Ablation (FLA) for BPH Active Treatment
Number analyzed (Participants) | 10
units on a scale | -17.5 (4.3)

2. Primary Outcome: International Prostate Symptom Score (IPSS) Quality of Life (QoL) Question Change
Description: The IPSS QoL question asks patients to rate how they would feel if they were to spend the rest of their lives with their urinary condition just the way it is now, from 0 ("delighted") to 6 ("terrible")
Time Frame: From baseline to 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Focal Laser Ablation (FLA) for BPH Active Treatment
Number analyzed (Participants) | 10
units on a scale | -3.4 (0.8)

3. Primary Outcome: BPH Impact Index Change
Description: This is another survey which rates lower urinary tract symptoms from 0 (none) to 13 (severe)
Time Frame: From baseline to 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Focal Laser Ablation (FLA) for BPH Active Treatment
Number analyzed (Participants) | 10
units on a scale | -6.9 (2.1)

4. Primary Outcome: Sexual Health Inventory of Men (SHIM) Score Change
Description: This survey rates erectile function from 0 (no function) to 25 (full function)
Time Frame: From baseline to 2 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Focal Laser Ablation (FLA) for BPH Active Treatment
Number analyzed (Participants) | 10
score on a scale | 1.9 (2.7)

5. Primary Outcome: Number of Adverse Events
Description: We asked patients to self-report adverse events.
Time Frame: Continuous until completion of the study at 2 years
Population: Two patients experienced urinary tract infections, two patients developed retrograde ejaculation, and one patient had urinary retention after foley catheter removal, requiring catheter replacement and maintenance for 1 week. All adverse events were considered mild using the Society of Interventional Radiology Adverse Events Classification System.
Measure: Count of Participants; unit: Participants
Arm/Group | FLA for BPH Active Treatment
Number analyzed (Participants) | 10
Participants | 4

6. Primary Outcome: International Prostate Symptom Score (IPSS) Change
Description: The IPSS survey rates lower urinary tract symptom severity from 0 (none) to 35 (severe).
Time Frame: From baseline to 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Focal Laser Ablation (FLA) for BPH Active Treatment
Number analyzed (Participants) | 10
units on a scale | -18.4 (4.2)

7. Primary Outcome: International Prostate Symptom Score (IPSS) Quality of Life (QoL) Question Change
Description: as for outcome 2
Time Frame: From baseline to 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Focal Laser Ablation (FLA) for BPH Active Treatment
Number analyzed (Participants) | 10
units on a scale | -3.1 (1.0)

8. Primary Outcome: BPH Impact Index Change
Description: This is another survey which rates lower urinary tract symptoms from 0 (none) to 13 (severe)
Time Frame: From baseline to 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Focal Laser Ablation (FLA) for BPH Active Treatment
Number analyzed (Participants) | 10
units on a scale | -7.4 (2.3)

9. Primary Outcome: Sexual Health Inventory of Men (SHIM) Score Change
Description: This survey rates erectile function from 0 (no function) to 25 (full function)
Time Frame: From baseline to 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Focal Laser Ablation (FLA) for BPH Active Treatment
Number analyzed (Participants) | 10
units on a scale | 1.1 (3.1)

10. Primary Outcome: International Prostate Symptom Score (IPSS) Change
Description: The IPSS survey rates lower urinary tract symptom severity from 0 (none) to 35 (severe).
Time Frame: From baseline to 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Focal Laser Ablation (FLA) for BPH Active Treatment
Number analyzed (Participants) | 10
units on a scale | -17.5 (4.1)

11. Primary Outcome: International Prostate Symptom Score (IPSS) Quality of Life (QoL) Question Change
Description: as for outcome 2
Time Frame: From baseline to 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Focal Laser Ablation (FLA) for BPH Active Treatment
Number analyzed (Participants) | 10
units on a scale | -3.2 (1.2)

12. Primary Outcome: BPH Impact Index Change
Description: This is another survey which rates lower urinary tract symptoms from 0 (none) to 13 (severe)
Time Frame: From baseline to 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Focal Laser Ablation (FLA) for BPH Active Treatment
Number analyzed (Participants) | 10
units on a scale | -6.7 (2.3)

13. Primary Outcome: Sexual Health Inventory of Men (SHIM) Score Change
Description: This survey rates erectile function from 0 (no function) to 25 (full function)
Time Frame: From baseline to 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Focal Laser Ablation (FLA) for BPH Active Treatment
Number analyzed (Participants) | 10
units on a scale | 0.8 (3.3)

14. Primary Outcome: International Prostate Symptom Score (IPSS) Change
Description: The IPSS survey rates lower urinary tract symptom severity from 0 (none) to 35 (severe).
Time Frame: From baseline to 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Focal Laser Ablation (FLA) for BPH Active Treatment
Number analyzed (Participants) | 9
units on a scale | -20.1 (5.8)

15. Primary Outcome: International Prostate Symptom Score (IPSS) Quality of Life (QoL) Question Change
Description: as for outcome 2
Time Frame: From baseline to 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Focal Laser Ablation (FLA) for BPH Active Treatment
Number analyzed (Participants) | 9
units on a scale | -3.7 (1.3)

16. Primary Outcome: BPH Impact Index Change
Description: This is another survey which rates lower urinary tract symptoms from 0 (none) to 13 (severe)
Time Frame: From baseline to 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Focal Laser Ablation (FLA) for BPH Active Treatment
Number analyzed (Participants) | 9
units on a scale | -7.7 (2.0)

17. Primary Outcome: Sexual Health Inventory of Men (SHIM) Score Change
Description: This survey rates erectile function from 0 (no function) to 25 (full function)
Time Frame: From baseline to 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Focal Laser Ablation (FLA) for BPH Active Treatment
Number analyzed (Participants) | 9
units on a scale | 2.8 (3.3)

ADVERSE EVENTS:
Time Frame: 2 years
Description: The patients were instructed to self-report their adverse events to us.
Arm/Group | FLA for BPH Active Treatment
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FLA for BPH Active Treatment (N=10)
Urinary tract infection (UTI) (Renal and urinary disorders) | 2 (2) — Both reported UTIs were lower urinary tract infections, likely related to the foley catheter
Retrograde ejaculation (Reproductive system and breast disorders) | 2 (2) — Retrograde ejaculation occurs when semen enters the bladder instead of emerging through the penis during orgasm.
Urinary retention (Renal and urinary disorders) | 1 (1) — Inability to urinate without difficulty after removal of foley catheter.

LIMITATIONS AND CAVEATS:
One patient dropped out after 6 month because his symptoms returned and he underwent a TURP.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-07): https://cdn.clinicaltrials.gov/large-docs/44/NCT03131544/Prot_SAP_000.pdf